CLINICAL TRIAL: NCT00890396
Title: Pediatric Hydroxyurea Phase III Clinical Trial (BABY HUG) Follow-up Study
Brief Title: Long-Term Effects of Hydroxyurea in Children With Sickle Cell Anemia (The BABY HUG Follow-up Study)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 647; N01HB07160 (NIH)
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2009-07

CONDITIONS: Anemia, Sickle Cell
Keywords: Sickle Cell Anemia; Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Stored blood and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Active Follow-up: An active follow-up involved the performance of many of the laboratory tests and procedures done during BABY HUG clinical trials study. These included, but not limited to, serial laboratory parameters that were not part of routine clinical care such as Hgb F levels, pitted cell count, Howell-Jolly Body determination, a liver-spleen scan, diethylenetriaminepentaacetic acid (DTPA) glomerular filtration rate (GFR) measurement, creatinine clearance, Cystatin C, urine concentrating ability, transcranial Doppler, and neuropsychological testing.
  Interventions: Drug: Hydroxyurea
- Passive Follow-up: A passive follow-up involved the abstraction of clinical data from the medical record. Results of physical examinations and laboratory tests performed as part of routine clinical care were recorded.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Parents and child's doctor may plan to use or not to use hydroxyurea.

SUMMARY:
Sickle cell anemia (SCA) is an inherited blood disorder that can cause organ damage. The BABY HUG study is evaluating the use of the medication hydroxyurea at preventing organ damage in children with SCA. The purpose of this follow-up study is to evaluate the long-term effects of hydroxyurea in children who have participated in the BABY HUG study.

DETAILED DESCRIPTION:
SCA is an inherited blood disorder in which the body makes sickle-shaped red blood cells that contain abnormal hemoglobin. The sickled cells block blood flow in the vessels that lead to limbs and organs. This can cause pain, serious infections, and organ damage. The BABY HUG study (NCT00006400) is examining whether the medication hydroxyurea can prevent organ damage, especially in the spleen and kidneys, in children with SCA. This study is a follow-up study to the BABY HUG study and will enroll children who have participated in the BABY HUG study. The purpose of this study is to examine the long-term effects of using hydroxyurea as a treatment for SCA, including both the risks and benefits. Study researchers will also investigate the optimal age to begin treatment with hydroxyurea in children with SCA.

This study will enroll children between 2 and 7 years old who participated in the BABY HUG study. Hydroxyurea will not be provided to participants as part of this study, but participants may receive the medication from their own doctors. Parents of participants can choose for their child to participate in this study in one of two ways-by enrolling in either a passive follow-up group or an active follow-up group. For participants in the passive follow-up group, study researchers will review participants' medical records every 6 months, in addition to reviewing brain ultrasound tests and computed tomography (CT) or magnetic resonance imaging (MRI) scans, if completed. Participants will have a blood and urine collection at baseline and Year 4 (or at the end of the study, whichever comes first). Participants in the active follow-up group will take part in the same study procedures as participants in the passive follow-up group. In addition, at Year 2, participants in this group will undergo an additional blood and urine collection, a scanning procedure to obtain images of the liver and spleen, a kidney test, neuropsychological testing, and an ultrasound imaging test to evaluate liver and spleen size.

ELIGIBILITY:
Inclusion Criteria:

* All children who completed at least 18 months of follow-up visits in the initial BABY HUG study
* Children from the initial BABY HUG study who are on a chronic transfusion program or who are recipients of a bone marrow transplant

Exclusion Criteria:

* Any child who was not enrolled in the initial BABY HUG study for at least 18 months

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from the initial BABY HUG study who agree to participate in this follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Assmann, PhD, Principal Investigator — New England Research Institutes, Watertown, MA
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Howard University College of Medicine, Washington D.C., District of Columbia
  - University of Miami School of Medicine, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Children's Hospital of Michigan/Wayne State University, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Downstate Medical Center, Brooklyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Drexel University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects that were eligible for enrollment included all children who have completed at least 18 months of the BABY HUG Treatment Study.
Pre-assignment Details: Parents and the participants' health care providers, who had not yet been informed of the BABY HUG randomized treatment, selected open label hydroxyurea (HU) treatment or standard care (SC).
Groups:
- Active: An active follow-up involved the performance of many of the laboratory tests and procedures done during BABY HUG clinical trials study. These included, but not limited to, serial laboratory parameters that were not part of routine clinical care such as Hgb F levels, pitted cell count, Howell-Jolly Body determination, a liver-spleen scan, diethylenetriaminepentaacetic acid (DTPA) glomerular filtration rate (GFR) measurement, creatinine clearance, Cystatin C, urine concentrating ability, transcranial Doppler, and neuropsychological testing.
- Passive: A passive follow-up involved the abstraction of clinical data from the medical record. Results of physical examinations and laboratory tests performed as part of routine clinical care were recorded.
Period: Overall Study
Arm/Group | Active | Passive
Started | 127 | 36
Completed | 122 | 34
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active: An active follow-up involved the performance of many of the laboratory tests and procedures done during BABY HUG clinical trials study. These included, but not limited to, serial laboratory parameters that were not part of routine clinical care such as Hgb F levels, pitted cell count, Howell-Jolly Body determination, a liver-spleen scan, DTPA GFR measurement, creatinine clearance, Cystatin C, urine concentrating ability, transcranial Doppler, and neuropsychological testing. Patients could be on or off hydroxyurea at the start of Follow-Up Study I, and could change treatment during the study.
- Passive: A passive follow-up involved the abstraction of clinical data from the medical record. Results of physical examinations and laboratory tests performed as part of routine clinical care were recorded. Patients could be on or off hydroxyurea at the start of Follow-Up Study I, and could change treatment during the study.
- Total: Total of all reporting groups
Arm/Group | Active | Passive | Total
Number analyzed (Participants) | 127 | 36 | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 127 | 36 | 163
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.41 (1.12) | 4.65 (1.25) | 4.46 (1.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 25 | 93
  Male | 59 | 11 | 70
Region of Enrollment [Number; unit: participants]
  United States | 127 | 36 | 163

OUTCOME MEASURES:

1. Primary Outcome: Change in Qualitative Spleen Function From Randomized Control Trial Baseline Measurement - Compared Between Children Randomized to Hydroxyurea vs Placebo
Description: The change in splenic function from the randomized control trial baseline measurement was one of the primary outcomes. The change in splenic function (worse vs not-worse) was compared between the randomized treatment groups (hydroxyurea vs placebo). The change in splenic function from baseline to 48 months was defined as worse if it changed from normal to decreased or absent, or decreased to absent; and not worse if it changed from decreased to decreased, normal to normal, decreased to normal, absent to absent, or absent to decreased.
Time Frame: 48 Months from the date of randomization
Population: All subjects who had 48 month and baseline spleen function measurement.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized to Hydroxyurea: Subjects randomized to Hydroxyurea in the randomized phase III clinical trial.
- Randomized to Placebo: Subjects randomized to Placebo in the randomized phase III clinical trial.
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
Number analyzed (Participants) | 60 | 49
Participants
  Splenic function - worse from baseline | 16 | 15
  Splenic function - not worse from baseline | 44 | 34
Statistical Analysis 1: Comparison: Randomized to Hydroxyurea vs Randomized to Placebo; The primary analysis compared the frequency of worsening spleen function (from normal to decreased or absent, or from decreased to absent); Test type: Superiority; p = 0.67, Fisher Exact

2. Primary Outcome: Change in Qualitative Spleen Function From Randomized Control Trial Baseline Measurement - Compared Between Children on Hydroxyurea vs Off Hydroxyurea at Study Visit
Description: The change in splenic function from the randomized control trial baseline measurement was one of the primary outcomes.The change in splenic function (worse vs not-worse) was compared between children who were known to be on hydroxyurea vs. off hydroxyurea at the time of the visit. The change in splenic function from baseline to 48 months was defined as worse if it changed from normal to decreased or absent, or decreased to absent; and not worse if it changed from decreased to decreased, normal to normal, decreased to normal, absent to absent, or absent to decreased.
Time Frame: 48 Months from the date of randomization
Population: All subjects who were known to be on hydroxyurea vs. off hydroxyurea at the 48 month visit, and had 48 month and baseline spleen function measurement.
Measure: Count of Participants; unit: Participants
Groups:
- On Hydroxyurea at the Time of Visit: Subjects who were on hydroxyurea at the time of study visit
- Off Hydroxyurea at the Time of Visit: Subjects who were off hydroxyurea at the time of study visit
Arm/Group | On Hydroxyurea at the Time of Visit | Off Hydroxyurea at the Time of Visit
Number analyzed (Participants) | 88 | 18
Participants
  Splenic function - worse from baseline | 26 | 5
  Splenic function - not worse from baseline | 62 | 13
Statistical Analysis 1: Comparison: On Hydroxyurea at the Time of Visit vs Off Hydroxyurea at the Time of Visit; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.99, Fisher Exact

3. Primary Outcome: Change in the Percentage of Pitted Cell From Randomized Control Trial Baseline Measurement - Compared Between Children Randomized to Hydroxyurea vs Placebo
Description: The change in the percentage of pitted cell from randomized control trial baseline measurement was one of the primary outcomes. The change in the percentage of pitted cell was compared between the randomized treatment groups (hydroxyurea vs placebo).
Time Frame: 48 Months from the date of randomization
Population: All subjects who had 48 month and baseline pitted cell measurements.
Measure: Median (Inter-Quartile Range); unit: Percentage of pitted cell
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
Number analyzed (Participants) | 59 | 49
Percentage of pitted cell | -1.70 [-5.70 to 0.00] | -1.00 [-3.40 to -0.10]
Statistical Analysis 1: Comparison: Randomized to Hydroxyurea vs Randomized to Placebo; Kruskal-Wallis test was used to test if there were a statistically significant difference between the two treatment groups; Test type: Superiority; p = 0.61, Kruskal-Wallis

4. Primary Outcome: Change in the Percentage of Pitted Cell From Randomized Control Trial Baseline Measurement - Compared Between Children Randomized to Hydroxyurea vs Placebo
Description: as for outcome 3
Time Frame: 72 Months from the date of randomization
Population: All subjects who had 72 month and baseline pitted cell measurements.
Measure: Median (Inter-Quartile Range); unit: Percentage of pitted cell
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
Number analyzed (Participants) | 70 | 64
Percentage of pitted cell | -1.55 [-5.70 to -0.30] | -1.40 [-4.75 to -0.35]
Statistical Analysis 1: Comparison: Randomized to Hydroxyurea vs Randomized to Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.78, Kruskal-Wallis

5. Primary Outcome: Change in the Percentage of Pitted Cell From Randomized Control Trial Baseline Measurement - Compared Between Children on Hydroxyurea vs Off Hydroxyurea at Study Visit
Description: The change in the percentage of pitted cell from the randomized control trial baseline measurement was one of the primary outcomes. The change in the percentage of pitted cell was compared between children who were known to be on hydroxyurea vs. off hydroxyurea at the time of the visit.
Time Frame: 48 Months from the date of randomization
Population: All subjects who were known to be on hydroxyurea vs. off hydroxyurea at the 48 month visit, and had 48 month and baseline pitted cell measurements.
Measure: Median (Inter-Quartile Range); unit: Percentage of pitted cell
Arm/Group | On Hydroxyurea at the Time of Visit | Off Hydroxyurea at the Time of Visit
Number analyzed (Participants) | 91 | 15
Percentage of pitted cell | -1.40 [-5.00 to -0.10] | -0.60 [-3.60 to 0.70]
Statistical Analysis 1: Comparison: On Hydroxyurea at the Time of Visit vs Off Hydroxyurea at the Time of Visit; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.80, Kruskal-Wallis

6. Primary Outcome: Change in the Percentage of Pitted Cell From Randomized Control Trial Baseline Measurement - Compared Between Children on Hydroxyurea vs Off Hydroxyurea at Study Visit
Description: as for outcome 5
Time Frame: 72 Months from the date of randomization
Population: All subjects who were known to be on hydroxyurea vs. off hydroxyurea at the 72 month visit, and had 72 month and baseline pitted cell measurements.
Measure: Median (Inter-Quartile Range); unit: Percentage of pitted cell
Arm/Group | On Hydroxyurea at the Time of Visit | Off Hydroxyurea at the Time of Visit
Number analyzed (Participants) | 104 | 27
Percentage of pitted cell | -1.30 [-4.65 to -0.25] | -1.70 [-11.10 to -0.50]
Statistical Analysis 1: Comparison: On Hydroxyurea at the Time of Visit vs Off Hydroxyurea at the Time of Visit; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.11, Kruskal-Wallis

7. Primary Outcome: Change in Howell-Jolly Bodies (HJB) From Randomized Control Trial Baseline Measurement - Compared Between Children Randomized to Hydroxyurea vs Placebo
Description: The change in Howell-Jolly Bodies from randomized control trial baseline measurement was one of the primary outcomes. The change in Howell-Jolly Bodies was compared between the randomized treatment groups (hydroxyurea vs placebo).
Time Frame: 48 Months from the date of randomization
Population: All subjects who had 48 month and baseline Howell-Jolly Bodies measurements.
Measure: Median (Inter-Quartile Range); unit: Number of HJB per 10⁶ red blood cell
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
Number analyzed (Participants) | 52 | 40
Number of HJB per 10⁶ red blood cell | 1626.25 [921.00 to 2316.50] | 1553.00 [189.00 to 2231.50]
Statistical Analysis 1: Comparison: Randomized to Hydroxyurea vs Randomized to Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.85, Kruskal-Wallis

8. Primary Outcome: Change in Howell-Jolly Bodies (HJB) From Randomized Control Trial Baseline Measurement - Compared Between Children Randomized to Hydroxyurea vs Placebo
Description: as for outcome 7
Time Frame: 72 Months from the date of randomization
Population: All subjects who had 72 month and baseline Howell-Jolly Bodies measurements.
Measure: Median (Inter-Quartile Range); unit: Number of HJB per 10⁶ red blood cell
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
Number analyzed (Participants) | 22 | 20
Number of HJB per 10⁶ red blood cell | 1847.50 [1270.00 to 2474.00] | 1906.50 [721.50 to 2679.50]
Statistical Analysis 1: Comparison: Randomized to Hydroxyurea vs Randomized to Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.95, Kruskal-Wallis

9. Primary Outcome: Change in Howell-Jolly Bodies (HJB) From Randomized Control Trial Baseline Measurement - Compared Between Children on Hydroxyurea vs Off Hydroxyurea at Study Visit
Description: The change in Howell-Jolly Bodies from the randomized control trial baseline measurement was one of the primary outcomes. The change in Howell-Jolly Bodies was compared between children who were known to be on hydroxyurea vs. off hydroxyurea at the time of the visit.
Time Frame: 48 Months from the date of randomization
Population: All subjects who were known to be on hydroxyurea vs. off hydroxyurea at the 48 month visit, and had 48 month and baseline Howell-Jolly Bodies measurements.
Measure: Median (Inter-Quartile Range); unit: Number of HJB per 10⁶ red blood cell
Arm/Group | On Hydroxyurea at the Time of Visit | Off Hydroxyurea at the Time of Visit
Number analyzed (Participants) | 79 | 11
Number of HJB per 10⁶ red blood cell | 1661.00 [796.00 to 2325.00] | 1510.00 [594.00 to 1875.00]
Statistical Analysis 1: Comparison: On Hydroxyurea at the Time of Visit vs Off Hydroxyurea at the Time of Visit; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.40, Kruskal-Wallis

10. Primary Outcome: Change in Howell-Jolly Bodies From Randomized Control Trial Baseline Measurement - Compared Between Children on Hydroxyurea vs Off Hydroxyurea at Study Visit
Description: The change in Howell-Jolly Bodies (HJB) from the randomized control trial baseline measurement was one of the primary outcomes. The change in Howell-Jolly Bodies was compared between children who were known to be on hydroxyurea vs. off hydroxyurea at the time of the visit.
Time Frame: 72 Months from the date of randomization
Population: All subjects who were known to be on hydroxyurea vs. off hydroxyurea at the 72 month visit, and had 72 month and baseline Howell-Jolly Bodies measurements.
Measure: Median (Inter-Quartile Range); unit: Number of HJB per 10⁶ red blood cell
Arm/Group | On Hydroxyurea at the Time of Visit | Off Hydroxyurea at the Time of Visit
Number analyzed (Participants) | 29 | 12
Number of HJB per 10⁶ red blood cell | 1972.00 [1270.00 to 2530.00] | 1500.50 [622.50 to 2043.50]
Statistical Analysis 1: Comparison: On Hydroxyurea at the Time of Visit vs Off Hydroxyurea at the Time of Visit; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.11, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: The date of consent to follow-up study I (FUS-I) through end of FUS-I, up to 2 years
Description: Serious adverse event (SAE) were Death, Life-threatening event, Prolonged hospitalization (greater than 7 days), Splenic sequestration crisis, Stroke / transient ischemic attack (TIA), Acute chest syndrome, or ICU admissions, and occurred during the first 5 days following performance of an active assessment study.
Arm/Group | Randomized to Hydroxyurea | Randomized to Placebo
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/79
Serious Adverse Events (participants affected / at risk) | 1/84 | 1/79
Other Adverse Events (participants affected / at risk) | 0/84 | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized to Hydroxyurea (N=84) | Randomized to Placebo (N=79)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Most children used hydroxyurea (HU) for at least part of the FUS-I observation period. This may dilute any effect of randomized group.

Most children were on HU at the specified time points, which reduces power to compare on/off HU.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: BABY HUG Randomized Control Trial (2009-08-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT00890396/Prot_SAP_000.pdf
  • Informed Consent Form: BABY HUG Randomized Control Trial (2006-10-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT00890396/ICF_001.pdf
  • Informed Consent Form: BABY HUG Follow-up Study I (2006-11-10): https://cdn.clinicaltrials.gov/large-docs/96/NCT00890396/ICF_002.pdf
  • Study Protocol and Statistical Analysis Plan: BABY HUG Follow-up Study I (2010-01-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT00890396/Prot_SAP_003.pdf